CLINICAL TRIAL: NCT00806819
Title: Multicenter, Randomized, Double-blind, Phase III Trial to Investigate the Efficacy and Safety of Oral BIBF 1120 Plus Standard Pemetrexed Therapy Compared to Placebo Plus Standard Pemetrexed Therapy in Patients With Stage IIIB/IV or Recurrent Non Small Cell Lung Cancer After Failure of First Line Chemotherapy
Brief Title: Lume Lung 2 : BIBF 1120 Plus Pemetrexed Compared to Placebo Plus Pemetrexed in 2nd Line Nonsquamous NSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.14; 2008-002072-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nintedanib; Pemetrexed; Vitamin B 12; Dexamethasone; Folic Acid

ARMS (5):
- nintedanib (BIBF1120) plus pemetrexed (Experimental): nintedanib (BIBF1120) along with standard therapy of pemetrexed
  Interventions: Drug: Nintedanib (BIBF1120); Drug: B12; Drug: dexamethasone (or corticosteroid equivalent); Drug: Folic Acid; Drug: Pemetrexed
- Placebo plus pemetrexed (Placebo Comparator): Pemetrexed standard therapy
  Interventions: Drug: pemetrexed; Drug: dexamethasone (or corticosteroid equivalent); Drug: B12; Drug: placebo; Drug: Folic Acid
- nintedanib (BIBF1120) monotherapy (Experimental): nintedanib (BIBF1120) monotherapy only for patients who discontinue pemetrexed
  Interventions: Drug: Nintedanib (BIBF1120)
- pemetrexed monotherapy (Active Comparator): pemetrexed monotherapy only for patients who discontinue nintedanib (BIBF1120) or placebo
  Interventions: Drug: Pemetrexed; Drug: B12; Drug: dexamethasone (or corticosteroid equivalent); Drug: Folic Acid
- placebo monotherapy (Placebo Comparator): placebo monotherapy only for patients who discontinue pemetrexed
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Nintedanib (BIBF1120) — starting dose of 200 mg bid taken daily except on the day of pemetrexed infusion . The dose can be reduced to 150 bid and then to 100 mg bid.
  Arms: nintedanib (BIBF1120) plus pemetrexed
Drug: Pemetrexed — 500 mg/metre squared administered as an intravenous infusion over 10 minutes on Day 1 of each 21 day cycle.
  Arms: pemetrexed monotherapy
Drug: pemetrexed — 500 mg/metre squared administered as an intravenous infusion over 10 minutes on Day 1 of each 21 day cycle.
  Arms: Placebo plus pemetrexed
Drug: B12 — 1000 ug IM injection starting a week before first pemetrexed infusion and every 9 weeks thereafter until discontinuation of pemetrexed
  Arms: pemetrexed monotherapy
Drug: dexamethasone (or corticosteroid equivalent) — 4 mg PO bid the day before, the day of and the day after each pemetrexed infusion
  Arms: pemetrexed monotherapy
Drug: placebo — starting dose of 200 mg bid taken daily except on the day of pemetrexed infusion . The dose can be reduced to 150 bid and then to 100 mg bid.
  Arms: placebo monotherapy
Drug: dexamethasone (or corticosteroid equivalent) — 4 mg PO bid the day before, the day of and the day after each pemetrexed infusion
  Arms: Placebo plus pemetrexed
Drug: B12 — 1000 ug IM injection starting a week before first pemetrexed infusion and every 9 weeks thereafter until discontinuation of pemetrexed
  Arms: nintedanib (BIBF1120) plus pemetrexed
Drug: Folic Acid — 400 ug once daily starting 1-2 weeks prior to the first dose of pemetrexed and continuing for at least 3 weeks after stopping pemetrexed.
  Arms: pemetrexed monotherapy
Drug: B12 — 1000 ug IM injection starting a week before first pemetrexed infusion and every 9 weeks thereafter until discontinuation of pemetrexed
  Arms: Placebo plus pemetrexed
Drug: dexamethasone (or corticosteroid equivalent) — 4 mg PO bid the day before, the day of and the day after each pemetrexed infusion
  Arms: nintedanib (BIBF1120) plus pemetrexed
Drug: Folic Acid — 400 ug once daily starting 1-2 weeks prior to the first dose of pemetrexed and continuing for at least 3 weeks after stopping pemetrexed.
  Arms: nintedanib (BIBF1120) plus pemetrexed
Drug: placebo — starting dose of 200 mg bid taken daily except on the day of pemetrexed infusion . The dose can be reduced to 150 bid and then to 100 mg bid.
  Arms: Placebo plus pemetrexed
Drug: Folic Acid — 400 ug once daily starting 1-2 weeks prior to the first dose of pemetrexed and continuing for at least 3 weeks after stopping pemetrexed.
  Arms: Placebo plus pemetrexed
Drug: Nintedanib (BIBF1120) — starting dose of 200 mg bid taken daily except on the day of pemetrexed infusion . The dose can be reduced to 150 bid and then to 100 mg bid.
  Arms: nintedanib (BIBF1120) monotherapy
Drug: Pemetrexed — 500 mg/metre squared administered as an intravenous infusion over 10 minutes on Day 1 of each 21 day cycle.
  Arms: nintedanib (BIBF1120) plus pemetrexed

SUMMARY:
The trial will be performed to evaluate if BIBF 1120 in combination with standard pemetrexed therapy is more effective than placebo (inactive capsule) plus standard pemetrexed therapy in patients with stage IIIB, IV or recurrent NSCLC. Safety information about BIBF1120/pemetrexed will be obtained.

ELIGIBILITY:
Inclusion criteria:

1. Male or female patient aged 18 years or older.
2. Histologically or cytologically confirmed Stage IIIB, IV (according to AJCC) or recurrent non small cell lung cancer (NSCLC) (non squamous histologies)
3. Relapse or failure of one first line chemotherapy (in the case of recurrent disease one additional prior regimen is allowed for adjuvant, neoadjuvant or neoadjuvant plus adjuvant therapy).
4. At least one target tumor lesion that has not been irradiated within the past three months and that can accurately be measured by magnetic resonance imaging (MRI) or computed tomography (CT) in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral CT.
5. Life expectancy of at least three months.
6. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
7. Patient has given written informed consent which must be consistent with the International Conference on Harmonization, Good Clinical Practice (ICH-GCP) and local legislation.

Exclusion criteria:

1. Previous therapy with other vascular endothelial growth factor (VEGF) inhibitors (other than bevacizumab) or pemetrexed for treatment of NSCLC
2. Treatment with other investigational drugs or treatment in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial
3. Chemotherapy, hormone therapy, immunotherapy with monoclonal antibodies, treatment with tyrosine kinase inhibitors, or radiotherapy (except for treatment of extremities) within the past four weeks prior to treatment with the trial drug, i.e., the minimum time elapsed since the last anticancer therapy and the first administration of BIBF 1120 must be four weeks
4. Inability to stop intake of NSAIDS (non steroidal anti inflammatory drugs) for several days
5. Active brain metastases (e.g. stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants). Dexamethasone therapy will be allowed if administered as stable dose for at least one month before randomisation)
6. Radiographic evidence of cavitary or necrotic tumors
7. Centrally located tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels
8. History of clinically significant haemoptysis within the past 3 months
9. Therapeutic anticoagulation
10. History of major thrombotic or clinically relevant major bleeding event in the past 6 months
11. Significant cardiovascular diseases (i.e., hypertension not controlled by medical therapy, unstable angina, history of myocardial infarction within the past 6 months,
12. Inadequate kidney, liver, blood clotting function
13. Inadequate blood count
14. Significant weight loss (> 10 %) within the past 6 weeks prior to treatment in the present trial
15. Current peripheral neuropathy greater than or equal to Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 except due to trauma
16. Pre-existing ascites (abdominal fluid collection) and/or clinically significant pleural effusion ( fluid collection between the lung and chest wall)
17. Major injuries and/or surgery within the past ten days prior to start of study drug
18. Incomplete wound healing
19. Active or chronic hepatitis C and/or B infection Additional exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2008-12; Primary Completion 2011-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (163):
- United States (40):
  - Boehringer Ingelheim Investigational Site, Downy, California
  - Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - Boehringer Ingelheim Investigational Site, Fullerton, California
  - Boehringer Ingelheim Investigational Site, Long Beach, California
  - Boehringer Ingelheim Investigational Site, Meriden, Connecticut
  - Boehringer Ingelheim Investigational Site, Aventura, Florida
  - Boehringer Ingelheim Investigational Site, Boynton Beach, Florida
  - Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - Boehringer Ingelheim Investigational Site, Miami, Florida
  - Boehringer Ingelheim Investigational Site, New Port Richey, Florida
  - Boehringer Ingelheim Investigational Site, Port Saint Lucie, Florida
  - Boehringer Ingelheim Investigational Site, Stuart, Florida
  - Boehringer Ingelheim Investigational Site, Galesburg, Illinois
  - Boehringer Ingelheim Investigational Site, Skokie, Illinois
  - Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - Boehringer Ingelheim Investigational Site, New Albany, Indiana
  - Boehringer Ingelheim Investigational Site, Witchita, Kansas
  - Boehringer Ingelheim Investigational Site, Ashland, Kentucky
  - Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - Boehringer Ingelheim Investigational Site, Burlington, Massachusetts
  - Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - Boehringer Ingelheim Investigational Site, Saint Louis Park, Minnesota
  - Boehringer Ingelheim Investigational Site, Grand Island, Nebraska
  - Boehringer Ingelheim Investigational Site, Farmington, New Mexico
  - Boehringer Ingelheim Investigational Site, Dunkirk, New York
  - Boehringer Ingelheim Investigational Site, Goshen, New York
  - Boehringer Ingelheim Investigational Site, Lake Success, New York
  - Boehringer Ingelheim Investigational Site, Nyack, New York
  - Boehringer Ingelheim Investigational Site, Asheville, North Carolina
  - Boehringer Ingelheim Investigational Site, Canton, Ohio
  - Boehringer Ingelheim Investigational Site, Sandusky, Ohio
  - Boehringer Ingelheim Investigational Site, Ephrata, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Langhorne, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Germantown, Tennessee
  - Boehringer Ingelheim Investigational Site, Amarillo, Texas
  - Boehringer Ingelheim Investigational Site, Seattle, Washington
  - Boehringer Ingelheim Investigational Site, Spokane, Washington
  - Boehringer Ingelheim Investigational Site, Madison, Wisconsin
  - Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Argentina (6):
  - Boehringer Ingelheim Investigational Site, Bs. As. Codigo Buenos Aires
  - Boehringer Ingelheim Investigational Site, Córdoba
  - Boehringer Ingelheim Investigational Site, Pergamino
  - Boehringer Ingelheim Investigational Site, Quilmes Buenos Aires
  - Boehringer Ingelheim Investigational Site, Rosario, Santa Fe
  - Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
- Australia (7):
  - Boehringer Ingelheim Investigational Site, Sydney, New South Wales
  - Boehringer Ingelheim Investigational Site, Brisbane, Queensland
  - Boehringer Ingelheim Investigational Site, Adelaide, South Australia
  - Boehringer Ingelheim Investigational Site, Toorak Gardens, South Australia
  - Boehringer Ingelheim Investigational Site, Melbourne, Victoria
  - Boehringer Ingelheim Investigational Site, Perth, Western Australia
  - Boehringer Ingelheim Investigational Site, Sydney
- Bosnia and Herzegovina (2):
  - Boehringer Ingelheim Investigational Site, Banja Luka
  - Boehringer Ingelheim Investigational Site, Sarajevo
- Brazil (20):
  - Boehringer Ingelheim Investigational Site, Belo Horizonte
  - Boehringer Ingelheim Investigational Site, Belo Horizonte,Minas Gerais
  - Boehringer Ingelheim Investigational Site, Cachoeira Do Itapemirim-ES
  - Boehringer Ingelheim Investigational Site, Campinas SP
  - Boehringer Ingelheim Investigational Site, Caxias do Sul
  - Boehringer Ingelheim Investigational Site, Curitiba
  - Boehringer Ingelheim Investigational Site, Florianópolis
  - Boehringer Ingelheim Investigational Site, Goiania Goias
  - Boehringer Ingelheim Investigational Site, Ijuí
  - Boehringer Ingelheim Investigational Site, Itajaí
  - Boehringer Ingelheim Investigational Site, Jau/SP
  - Boehringer Ingelheim Investigational Site, Londrina, Parana
  - Boehringer Ingelheim Investigational Site, Pelotas Rio Grande Do Sul
  - Boehringer Ingelheim Investigational Site, Porto Alegre
  - Boehringer Ingelheim Investigational Site, Rio de Janeiro
  - Boehringer Ingelheim Investigational Site, Salvador Bahia
  - Boehringer Ingelheim Investigational Site, Santo André
  - Boehringer Ingelheim Investigational Site, Sao Paulo - SP
  - Boehringer Ingelheim Investigational Site, São Paulo
  - Boehringer Ingelheim Investigational Site, Sorocaba Sao Paulo
- Canada (4):
  - Boehringer Ingelheim Investigational Site, Thunder Bay, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - Boehringer Ingelheim Investigational Site, Québec, Quebec
- Chile (4):
  - Boehringer Ingelheim Investigational Site, Jardin Del Mar, Renaca
  - Boehringer Ingelheim Investigational Site, Las Condes
  - Boehringer Ingelheim Investigational Site, Santiago
  - Boehringer Ingelheim Investigational Site, Temuco
- Boehringer Ingelheim Investigational Site, Monteria, Cordoba, Colombia
- Ecuador (2):
  - Boehringer Ingelheim Investigational Site, Cuenca
  - Boehringer Ingelheim Investigational Site, Quito
- Germany (6):
  - Boehringer Ingelheim Investigational Site, Augsburg
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Gauting
  - Boehringer Ingelheim Investigational Site, Halle
  - Boehringer Ingelheim Investigational Site, Hemer
  - Boehringer Ingelheim Investigational Site, München
- Boehringer Ingelheim Investigational Site, Hong Kong, Hong Kong
- Hungary (3):
  - Boehringer Ingelheim Investigational Site, Deszk
  - Boehringer Ingelheim Investigational Site, Nyíregyháza
  - Boehringer Ingelheim Investigational Site, Pécs
- Boehringer Ingelheim Investigational Site, Dublin, Ireland
- Latvia (3):
  - Boehringer Ingelheim Investigational Site, Daugavpils
  - Boehringer Ingelheim Investigational Site, Liepāja
  - Boehringer Ingelheim Investigational Site, Riga
- Malaysia (4):
  - Boehringer Ingelheim Investigational Site, George Town
  - Boehringer Ingelheim Investigational Site, Kota Kinabalu
  - Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - Boehringer Ingelheim Investigational Site, Kuching
- Mexico (2):
  - Boehringer Ingelheim Investigational Site, Chihuahua City
  - Boehringer Ingelheim Investigational Site, Morelia
- Boehringer Ingelheim Investigational Site, Chisinau, Moldova
- Boehringer Ingelheim Investigational Site, 's-Hertogenbosch, Netherlands
- New Zealand (4):
  - Boehringer Ingelheim Investigational Site, Auckland
  - Boehringer Ingelheim Investigational Site, Christchurch
  - Boehringer Ingelheim Investigational Site, Palmerston North
  - Boehringer Ingelheim Investigational Site, Wellington
- North Macedonia (2):
  - Boehringer Ingelheim Investigational Site, Bitola
  - Boehringer Ingelheim Investigational Site, Skopje
- Panama (2):
  - Boehringer Ingelheim Investigational Site, Carrasquilla Panama
  - Boehringer Ingelheim Investigational Site, Panama City
- Peru (3):
  - Boehringer Ingelheim Investigational Site, Arequipa
  - Boehringer Ingelheim Investigational Site, Cercado Arequipa
  - Boehringer Ingelheim Investigational Site, Lima
- Philippines (4):
  - Boehringer Ingelheim Investigational Site, Cebu
  - Boehringer Ingelheim Investigational Site, Davao City
  - Boehringer Ingelheim Investigational Site, Makati
  - Boehringer Ingelheim Investigational Site, Quezon
- Boehringer Ingelheim Investigational Site, Olsztyn, Poland
- Romania (6):
  - Boehringer Ingelheim Investigational Site, Baia Mare
  - Boehringer Ingelheim Investigational Site, Bucharest
  - Boehringer Ingelheim Investigational Site, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site, Iași
  - Boehringer Ingelheim Investigational Site, Onești
  - Boehringer Ingelheim Investigational Site, Timișoara
- Serbia (3):
  - Boehringer Ingelheim Investigational Site, Belgrade
  - Boehringer Ingelheim Investigational Site, Kamenitz
  - Boehringer Ingelheim Investigational Site, Niš
- South Korea (8):
  - Boehringer Ingelheim Investigational Site, Daegu
  - Boehringer Ingelheim Investigational Site, Daejoen
  - Boehringer Ingelheim Investigational Site, Gangdong-gu, Seoul
  - Boehringer Ingelheim Investigational Site, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site, Jeonbuk
  - Boehringer Ingelheim Investigational Site, Seochogu, Seoul
  - Boehringer Ingelheim Investigational Site, Seoul
  - Boehringer Ingelheim Investigational Site, Suwon
- Sweden (4):
  - Boehringer Ingelheim Investigational Site, Gävle
  - Boehringer Ingelheim Investigational Site, Stockholm
  - Boehringer Ingelheim Investigational Site, Umeå
  - Boehringer Ingelheim Investigational Site, Uppsala
- Taiwan (4):
  - Boehringer Ingelheim Investigational Site, Kaohsiung City
  - Boehringer Ingelheim Investigational Site, Taichung
  - Boehringer Ingelheim Investigational Site, Tainan
  - Boehringer Ingelheim Investigational Site, Taipei
- Thailand (2):
  - Boehringer Ingelheim Investigational Site, Bangkok
  - Boehringer Ingelheim Investigational Site, Chiang Mai
- Turkey (Türkiye) (7):
  - Boehringer Ingelheim Investigational Site, Ankara
  - Boehringer Ingelheim Investigational Site, Antalya
  - Boehringer Ingelheim Investigational Site, Aydin
  - Boehringer Ingelheim Investigational Site, Balcali-Adana
  - Boehringer Ingelheim Investigational Site, Diyarbakır
  - Boehringer Ingelheim Investigational Site, Gaziantep
  - Boehringer Ingelheim Investigational Site, Kocaeli
- Ukraine (5):
  - Boehringer Ingelheim Investigational Site, Chernihiv
  - Boehringer Ingelheim Investigational Site, Dnipropetrovks
  - Boehringer Ingelheim Investigational Site, Kharkiv
  - Boehringer Ingelheim Investigational Site, Uzhhorod
  - Boehringer Ingelheim Investigational Site, Vinnytsia

REFERENCES:
- [Derived] Lesaffre E, Edelman MJ, Hanna NH, Park K, Thatcher N, Willemsen S, Gaschler-Markefski B, Kaiser R, Manegold C. Statistical controversies in clinical research: futility analyses in oncology-lessons on potential pitfalls from a randomized controlled trial. Ann Oncol. 2017 Jul 1;28(7):1419-1426. doi: 10.1093/annonc/mdx042. PMID 28184431

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 patients at one investigator site were excluded from the enrollment count because of site non-compliance.
Groups:
- Nintedanib Plus Pemetrexed: Nintedanib 200 mg twice daily administered orally in a form of a soft gelatin capsule on day2 to 21 of each 21-day treatment course plus pemetrexed 500 mg/m2 on Day1 of each 21-day treatment course administered via intravenous infusion. If required the dose of nitedanib could be redused to 150 mg twice daily (b.i.d.) or 100 mg b.i.d. and two dose reductions for pemetrexed were allowed (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
- Placebo Plus Pemetrexed: Placebo soft gelatin capsule matching that of nintedanib 2 times daily on day 2 to 21 of each 21-day treatment course administered orally plus pemetrexed 500 mg/m2 on Day 1 of each 21-day treatment course administered via intravenous infusion. If required two dose reductions for pemetrexed were allowed (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
Period: Overall Study
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Started | 353 (randomised patients) | 360 (randomised patients)
Completed | 7 (On-treatment at analysis DBL date (15 February 2013)) | 2 (On-treatment at analysis DBL date (15 February 2013))
Not Completed | 346 | 358
Not completed — progressive disease (modified RECIST ) | 217 | 216
Not completed — Worsening or AE of underlying disease | 18 | 25
Not completed — Other AE | 38 | 40
Not completed — Protocol Violation | 9 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 32 | 29
Not completed — Not treated | 6 | 3
Not completed — Reasons other than stated above | 25 | 41

BASELINE CHARACTERISTICS:
Population: Randomised set uncut (RS): all patients who were randomised whether patients had received study treatment or not. Patients were allocated to the treatment groups as randomised, regardless of the actual medication taken.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed | Total
Number analyzed (Participants) | 353 | 360 | 713
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (10.3) | 58.7 (10.9) | 59.0 (10.6)
Gender [Count of Participants; unit: Participants]
  Female | 158 | 152 | 310
  Male | 195 | 208 | 403

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by Central Independent Review
Description: Progression Free Survival (PFS) as assessed by central independent review according to the modified RECIST (version 1.0) criteria. Progression free survival (PFS) is defined as the duration of time from date of randomisation to date of progression or death (whatever occurs earlier).
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From randomisation until cut-off date 9 July 2012
Population: RS
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
months | 4.4 [2.3 to 9.5] | 3.6 [1.4 to 7.5]
Statistical Analysis 1: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; HR, CI and p-value obtained from the proportional hazards model stratified by baseline ECOG PS (0 vs 1), tumour histology (adenocarcinoma vs. non-adenocarcinoma), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Test type: Superiority or Other; p = 0.0435, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.70 to 0.99] — HR below 1 favors nintedanib

2. Secondary Outcome: Overall Survival (Key Secondary Endpoint)
Description: Overall Survival (OS) defined as the duration from randomisation to death (irrespective of the reason of death). Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From randomisation until data cut-off (15 February 2013), Up to 30 months
Population: RS
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
months | 12.0 [7.0 to 24.2] | 12.7 [5.4 to 24.0]
Statistical Analysis 1: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; HR, CI and p-value obtained from the prop. hazards model stratified by baseline ECOG PS (0 vs 1), tumour histology (adenocarcinoma vs non-adenocarcinoma), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Test type: Superiority or Other; p = 0.8940, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.85 to 1.21] — HR below 1 favors nintedanib

3. Secondary Outcome: Follow-up Analysis of Progression Free Survival (PFS) as Assessed by Central Independent Review
Description: Follow-up analysis was conducted at the time of overall survival analysis. Progression Free Survival (PFS) as assessed by central independent review according to the modified RECIST (version 1.0) criteria. Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From randomisation until data cut-off (15 February 2013), Up to 30 months
Population: RS
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
Months | 4.4 [2.3 to 9.5] | 3.4 [1.4 to 7.5]
Statistical Analysis 1: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0506, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.70 to 1.00] — HR below 1 favors nintedanib

4. Secondary Outcome: Follow-up Analysis of Progression Free Survival (PFS) as Assessed by Investigator
Description: Follow-up analysis was conducted at the time of overall survival analysis. Progression Free Survival (PFS) as assessed by investigator according to the modified RECIST (version 1.0) criteria. Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From randomisation until data cut-off (15 February 2013), Up to 30 months
Population: RS
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
Months | 5.3 [2.6 to 9.4] | 4.3 [1.9 to 8.3]
Statistical Analysis 1: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0865, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.73 to 1.02] — HR below 1 favors nintedanib

5. Secondary Outcome: Objective Tumor Response
Description: Confirmed objective response is defined as confirmed Complete Response (CR) and Partial Response (PR) and evaluated according to the modified RECIST criteria version 1.0. This endpoint was analysed based on the central independent reviewer as well as the investigator
Time Frame: From randomisation until data cut-off (15 February 2013), Up to 30 months
Population: Randomised Set
Measure: Number; unit: % of participants
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
% of participants
  Central independent reviewer | 9.1 | 8.3
  Investigator assessment | 15.0 | 13.3
Statistical Analysis 1: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; Analysis based on the central independent review; Test type: Superiority or Other; p = 0.7279, Regression, Logistic — Odds ratio and p-value are obtained from logistic regression model adjusted for baseline ECOG PS (0 vs 1); Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.65 to 1.85] — An odds ratio >1 indicates a benefit to nintedanib
Statistical Analysis 2: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; Analysis based on the investigator's assessment; Test type: Superiority or Other; p = 0.5180, Regression, Logistic — Odds ratio and p-value are obtained from logistic regression model adjusted for baseline ECOG PS (0 vs 1); Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.75 to 1.76] — An odds ratio >1 indicates a benefit to nintedanib

6. Secondary Outcome: Duration of Confirmed Objective Tumour Response
Description: The duration of objective response is the time from first documented (CR) or (PR) to the time of progression or death and evaluated according to the modified RECIST criteria version 1.0. Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
  This endpoint was analysed based on the central independent reviewer as well as the investigator.
Time Frame: From randomisation until data cut-off (15 February 2013), Up to 30 months
Population: RS
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
Months
  central independent reviewer (N=32, 30) | 6.9 [5.1 to 11.3] | 4.4 [3.3 to 8.9]
  Investigator assessment (N=53, 48) | 6.5 [4.4 to 12.7] | 7.2 [4.2 to 16.2]

7. Secondary Outcome: Time to Confirmed Objective Tumour Response
Description: Time to confirmed objective response is defined as time from randomisation to the date of first documented (CR) or (PR) and evaluated according to the modified RECIST criteria version 1.0. Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
  This endpoint was analysed based on the central independent reviewer as well as the investigator.
Time Frame: From randomisation until data cut-off (15 February 2013), Up to 30 months
Population: RS
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
Months
  Central independent review (N=32, 30) | 2.6 [1.4 to 4.0] | 2.7 [1.4 to 4.2]
  Investigator assessment (N=53, 48) | 2.6 [1.4 to 3.0] | 2.8 [1.4 to 3.1]

8. Secondary Outcome: Disease Control
Description: Disease control was defined as a best overall response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) and evaluated according to the modified RECIST criteria version 1.0.
  This endpoint was analysed based on the central independent reviewer as well as the investigator.
Time Frame: From randomisation until data cut-off (15 February 2013), Up to 30 months
Population: RS
Measure: Number; unit: % of participants
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
% of participants
  Central independent review (N=215, 192) | 60.9 | 53.3
  Investigator assessment (N=233, 217) | 66.0 | 60.3
Statistical Analysis 1: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; Analysis based on the central independent review; Test type: Superiority or Other; p = 0.0387, Regression, Logistic — Odds ratio and p-value are obtained from logistic regression model adjusted for baseline ECOG PS (0 vs 1); Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.02 to 1.85] — An odds ratio >1 indicates a benefit to nintedanib
Statistical Analysis 2: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; Analysis based on investigator's assessment; Test type: Superiority or Other; p = 0.1071, Regression, Logistic — Odds ratio and p-value are obtained from logistic regression model adjusted for baseline ECOG PS (0 vs 1); Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.95 to 1.75] — An odds ratio >1 indicates a benefit to nintedanib

9. Secondary Outcome: Duration of Disease Control
Description: The duration of disease control was defined as the time from randomisation to the date of disease progression or death (which ever occurs first) for patients with disease control. Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
  This endpoint was analysed based on the central independent reviewer as well as the investigator.
Time Frame: From randomisation until data cut-off (15 February 2013), Up to 30 months
Population: RS
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
Months
  Central independent review (N=215, 192) | 7.4 [4.3 to 11.2] | 6.8 [4.2 to 12.5]
  Investigator assessment (N=233, 217) | 6.9 [4.4 to 12.5] | 6.8 [4.4 to 11.1]

10. Secondary Outcome: Change From Baseline in Tumour Size
Description: Percentage change from baseline in tumour size is defined as decrease in the sum of the longest diameter of the target lesion. Presented means are in fact adjusted best means percentage changes generated from ANOVA model adjusted for baseline ECOG PS (0 vs. 1), tumour histology (adenocarcinoma vs. non-adenocarcinoma), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no) This endpoint was analysed based on the central independent reviewer as well as the investigator.
Time Frame: From randomisation until data cut-off (15 February 2013), Up to 30 months
Population: RS
Measure: Mean (95% Confidence Interval); unit: percentage of change in tumor size in mm
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
percentage of change in tumor size in mm
  Central independent review (N=298, 305) | -10.10 [-12.63 to -7.58] | -7.53 [-10.03 to -5.04]
  Investigator assessment (N=322, 325) | -15.60 [-18.75 to -12.46] | -11.28 [-14.42 to -8.15]
Statistical Analysis 1: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; Analysis based on the central independent review; Test type: Superiority or Other; p = 0.1558, ANOVA — P-value generated from ANOVA model adjusted for baseline ECOG PS (0 vs. 1), tumour histology (adenocarcinoma vs. non-adenocarcinoma), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no)
Statistical Analysis 2: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; Analysis based on the investigator's assessment; Test type: Superiority or Other; p = 0.0565, ANOVA — [p-value comment as in outcome 10, analysis 1]

11. Secondary Outcome: Clinical Improvement.
Description: Clinical improvement was defined as the time from randomisation to deterioration in body weight and/or Eastern Cooperative Oncology group performance score (ECOG PS) whichever occurred first.
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From randomisation until data cut-off (15 February 2013), Up to 30 months
Population: RS
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
Months | 7.2 [2.8 to 21.9] | 7.5 [1.8 to 24.2]
Statistical Analysis 1: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5068, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.74 to 1.16] — HR below 1 favors nintedanib

12. Secondary Outcome: Quality of Life (QoL)
Description: QoL was measured by standardised questionnaires (EQ-5D, EORTC QLQ-C30, EORTC QLQ-LC13). The EORTC QLQ-C30 comprises of 30 questions, using both multi-item scales and single-item measures. EORTC LC-13 comprises of 13 questions incorporating 1 multi-item scale and a series of single items. The following were the main points of interest: Time to deterioration of cough (QLQ-LC13 question 1), Time to deterioration of dyspnoea (QLQ-LC13, composite of questions 3 to 5), Time to deterioration of pain (QLQ- C30, composite of questions 9 and 19). Time to deterioration of cough, dyspnoea and pain was defined as the time to a 10-point increase from the baseline score.
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From randomisation until data cut-off (15 February 2013), Up to 30 months
Population: RS
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 353 | 360
Months
  Time to deterioration of cough | 6.0 [2.2 to 23.6] | 4.3 [1.4 to NA] — As only 43.9% of patients had a deterioration of cough by the cut-off date, the 75th percentile was not estimable.
  Time to deterioration of dyspnoea | 2.4 [0.9 to 6.4] | 2.0 [0.8 to 5.7]
  Time to deterioration of pain | 2.8 [1.2 to 7.0] | 2.7 [1.1 to 8.0]
Statistical Analysis 1: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; Analysis evaluating the time to deterioration of cough. HR, CI and p-value obtained from the prop. hazards model stratified by baseline ECOG PS (0 vs >=1), tumour histology (adenocarcinoma vs. non-adenocarcinoma), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Test type: Superiority or Other; p = 0.1181, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.66 to 1.05] — HR below 1 favors nintedanib
Statistical Analysis 2: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; Analysis evaluating the time to deterioration of dyspnoea. HR, CI and p-value obtained from the prop. hazards model stratified by baseline ECOG PS (0 vs >=1), tumour histology (adenocarcinoma vs. non-adenocarcinoma), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Test type: Superiority or Other; p = 0.4264, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.77 to 1.12] — HR below 1 favors nintedanib
Statistical Analysis 3: Comparison: Nintedanib Plus Pemetrexed vs Placebo Plus Pemetrexed; Analysis evaluating the time to deterioration of pain. HR, CI and p-value obtained from the prop. hazards model stratified by baseline ECOG PS (0 vs >= 1), tumour histology (adenocarcinoma vs. non-adenocarcinoma), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Test type: Superiority or Other; p = 0.8929, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.84 to 1.23] — HR below 1 favors nintedanib

13. Secondary Outcome: Dose Normalised Predose Plasma Concentration at Steady State (Cpre,ss,Norm) of Nintedanib and of Its Metabolites BIBF 1202 and BIBF 1202 Glucuronide
Description: Geometric mean of dose normalised predose plasma concentration (Cpre,ss,norm) of nintedanib and of its metabolites BIBF 1202 and BIBF 1202 glucuronide evaluated at steady state based on course 2 and 3. If only one value was available and valid, then this value was used for calculation of Cpre,ss,norm.
Time Frame: Before the administration of nintedanib or placebo and between a window of 30 mins to an hour after administration of trial drug during Course 2 and between 1 and 3 hours after administration of trial drug during Course 3
Population: Pharmacokinetic set- all patients in the treated set who were documented to have received at least 1 dose of nintedanib and who had at least 1 valid drug plasma concentration available
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Groups:
- Nintedanib 150 mg Bid Plus Pemetrexed: Nintedanib 150 mg twice daily administered orally in a form of a soft gelatin capsule plus pemetrexed 500 mg/m2 on Day 1 of each 21-day treatment course administered via intravenous infusion.
Arm/Group | Nintedanib Plus Pemetrexed | Nintedanib 150 mg Bid Plus Pemetrexed
Number analyzed (Participants) | 188 | 40
ng/mL/mg
  Nintedanib BIBF 1120 (N=188, 39) | 0.0883 (66.4) | 0.103 (72.9)
  Nintedanib BIBF 1202 (N=188, 40) | 0.131 (123) | 0.151 (125)
  Nintedanib BIBF 1202 glucuronide (N=184, 39) | 1.40 (169) | 1.72 (185)

14. Secondary Outcome: Incidence and Intensity of Adverse Events
Description: Incidence and intensity of adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. The worst CTCAE grade per patient is reported and MedDRA version 15.1 used.
  Serious signs and symptoms of progressive disease were reported as an adverse event in analysis of this endpoint.
Time Frame: From the first drug administration until 28 days after the last drug administration, up to 36 months
Population: Treated set uncut - all randomised patients who were documented to have taken at least 1 dose of study medication . Patients were allocated to the treatment groups according to the treatment actually received.
Measure: Number; unit: % of participants
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 347 | 357
% of participants
  CTCAE grade 1 | 4.9 | 9.2
  CTCAE grade 2 | 22.2 | 30.5
  CTCAE grade 3 | 46.1 | 34.5
  CTCAE grade 4 | 12.4 | 7.8
  CTCAE grade 5 | 9.8 | 12.0

ADVERSE EVENTS:
Time Frame: From the first drug administration until 28 days after the last drug administration, up to 36 months
Description: One patient in the nintedanib plus pemetrexed treatment arm reported a serious adverse event for which the preferred term was not yet coded until data cut-off (15 February 2013).
Arm/Group | Nintedanib Plus Pemetrexed | Placebo Plus Pemetrexed
Serious Adverse Events (participants affected / at risk) | 104/347 | 117/357
Other Adverse Events (participants affected / at risk) | 320/347 | 312/357
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib Plus Pemetrexed (N=347) | Placebo Plus Pemetrexed (N=357)
Anaemia (Blood and lymphatic system disorders) | 5 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 3
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 6
Asthenia (General disorders) | 0 | 3
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Disease progression (General disorders) | 2 | 1
Fatigue (General disorders) | 2 | 3
General physical health deterioration (General disorders) | 4 | 3
Mass (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 2
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 4
Spinal pain (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 2
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 1
Amoebiasis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 3
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Infectious peritonitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 2
Lymphangitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 1
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 11 | 16
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 1
Urosepsis (Infections and infestations) | 0 | 1
Chemical injury (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 2 | 1
Renal injury (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 3
Raynaud's phenomenon (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib Plus Pemetrexed (N=347) | Placebo Plus Pemetrexed (N=357)
Anaemia (Blood and lymphatic system disorders) | 26 | 23
Neutropenia (Blood and lymphatic system disorders) | 27 | 19
Lacrimation increased (Eye disorders) | 15 | 21
Abdominal pain (Gastrointestinal disorders) | 41 | 27
Abdominal pain upper (Gastrointestinal disorders) | 16 | 22
Constipation (Gastrointestinal disorders) | 50 | 65
Diarrhoea (Gastrointestinal disorders) | 118 | 54
Nausea (Gastrointestinal disorders) | 126 | 118
Stomatitis (Gastrointestinal disorders) | 27 | 21
Vomiting (Gastrointestinal disorders) | 84 | 68
Asthenia (General disorders) | 25 | 31
Chest pain (General disorders) | 31 | 29
Fatigue (General disorders) | 116 | 127
Oedema peripheral (General disorders) | 26 | 30
Pain (General disorders) | 17 | 21
Pyrexia (General disorders) | 36 | 42
Upper respiratory tract infection (Infections and infestations) | 21 | 20
Alanine aminotransferase increased (Investigations) | 149 | 87
Aspartate aminotransferase increased (Investigations) | 129 | 68
Blood alkaline phosphatase increased (Investigations) | 33 | 13
Haemoglobin decreased (Investigations) | 41 | 44
Neutrophil count decreased (Investigations) | 74 | 47
Platelet count decreased (Investigations) | 23 | 13
Weight decreased (Investigations) | 23 | 15
White blood cell count decreased (Investigations) | 57 | 38
Decreased appetite (Metabolism and nutrition disorders) | 97 | 89
Hyperglycaemia (Metabolism and nutrition disorders) | 24 | 28
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 36
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 27
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 16
Dizziness (Nervous system disorders) | 30 | 39
Headache (Nervous system disorders) | 44 | 47
Insomnia (Psychiatric disorders) | 29 | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 55 | 60
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45 | 70
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 | 12
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 29 | 29
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 33
Rash (Skin and subcutaneous tissue disorders) | 22 | 28

LIMITATIONS AND CAVEATS:
Recruitment for the study was stopped early based on the results of a pre defined futility analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.